CLINICAL TRIAL: NCT01962220
Title: Mother Infant Retention for Health: Evaluation of a Multicomponent Strategy to Link and Retain Newly Identified HIV-infected Pregnant Women and Their Infants Throughout the Antenatal and Post-partum Period
Brief Title: Mother Infant Retention for Health: MIR4Health
Acronym: MIR4HEALTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Kenya Ministry of Health (Other Government)
Responsible Party: Principal Investigator, Elaine J. Abrams, MD, Director Research Unit, ICAP, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAL5557; 1R01HD075163-01 (NIH)
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS; PMTCT; Pregnant Women; Kenya; Maternal Health
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention): Routine ANC, Delivery and Postpartum Care: All consenting women will receive routine ANC/Delivery and Postpartum care offered to pregnant women in Kenya as per national guidelines at the MCH of the respective facility.
  Routine PMTCT and HIV Care: All newly diagnosed HIV-infected pregnant women are enrolled into HIV care in the MCH and receive PMTCT/HIV care per Kenya national guidelines (Revised 2012 PMTCT Guidelines).
- Study Intervention for Retention (APFU) (Experimental): Participants randomized to the experimental arm of the study will receive routine antenatal and HIV services as described above per Kenya national guidelines. In addition each newly identified HIV-infected pregnant woman randomized to the experimental arm will be assigned an outreach worker/counselor (Mama Mshauri), who will perform numerous tasks described in the intervention. In addition to the Mama Mshauri, this arm will receive phone/SMS appointment reminders, and default patient tracking if participants miss an appointment.
  Interventions: Behavioral: Study Intervention for Retention (APFU)

INTERVENTIONS:
Behavioral: Study Intervention for Retention (APFU) — Each newly identified HIV-infected pregnant woman randomized to the experimental arm will be assigned an outreach worker/counselor (Mama Mshauri).
  Mama Mshauri tasks will include:
  * Immediately engaging the newly identified pregnant woman, providing individualized adherence and disclosure support, management of ART side effects, and helping the client navigate the health system.
  * Providing tailored individualized health education during home visits.
  Additional intervention components include:
  * Appointments and Reminders: SMS or telephone reminders 1 week and 3 days before appointments. Reinforcement of importance of follow-up during home visits and every contact.
  * Patient Tracking and Defaulter Tracing: Monthly visits and immediate calls/home visit if she misses an appointment.
  Arms: Study Intervention for Retention (APFU)

SUMMARY:
Linking HIV-infected pregnant women into prevention of mother to child transmission (PMTCT) services and keeping them in care is important in ensuring that both mother and infant beneﬁt from interventions that improve maternal health and decrease HIV transmission to infants. We propose an evaluation of strategies to link newly diagnosed HIV-infected women to care and keep them in care during pregnancy and after delivery in our study called MIR4HEALTH. The study will be conducted in Nyanza Province, Kenya. All participants will provide informed consent and will be randomized to receive the intervention, including individualized patient education, adherence support and phone call/Short Message Service (SMS) reminders for clinic appointments, or the standard of care (no additional intervention services).

DETAILED DESCRIPTION:
Mother Infant Retention for Health (MIR4HEALTH) is an innovative implementation science study focused on testing an effective multicomponent strategy to improve linkage and retention of newly identified HIV-infected pregnant women accessing maternal child health (MCH) services in Nyanza Province, Kenya. MIR4HEALTH is distinguished by several innovations including the recognition that newly identified HIV-infected pregnant woman are especially vulnerable to poor retention within PMTCT services and that both mother and child must be retained in care to ensure optimal health outcomes.

The study is a randomized trial to compare the effectiveness of a novel strategy using Active Patient Follow-Up (APFU) to the current standard of care (SOC) routinely provided for the retention of women and their exposed infants postpartum. The proposed APFU includes a package of evidence-based interventions including health education, provision of phone and short message service (SMS) appointment reminders, active tracking of patients for linkage and retention, and individualized retention and adherence support. Patients enrolled in the APFU intervention arm will complete three antenatal study visits after enrollment as well as two postnatal study visits with their infants at 6 weeks and 6 months postpartum. Laboratory blood specimens will be collected from mothers and infants at two separate visits to assess viral load and and drug levels. Additionally, all staff will be offered a chance to participate in an interview assessing the feasibility and acceptability of APFU.

Study participants will be recruited from various clinics in the Nyanza Province in Kenya. This study will enroll pregnant women who test positive for HIV during their first antenatal visit and have no prior HIV diagnosis. Upon live birth, the infants of participating women will also be included in the study. The study will enroll 214 newly-infected pregnant women, with 107 participants in the APFU arm (intervention) and 107 participants in the SOC arm. Infants born to women enrolled in the study will also be included so there will be a total of 214 mother-infant pairs, totaling 428 participants.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-infection according to two finger-prick rapid tests (both previously diagnosed and newly detected)
* Confirmed pregnancy by urine pregnancy test or clinical assessment
* Age 16 years or older
* Able to provide informed consent for research
* Fluent in Luo or English
* Own a cell phone or have access to one in their households
* Live born infants of women enrolled in the study

Exclusion Criteria:

* Patients who fail to meet any of the inclusion criteria will be excluded
* Significant obstetric condition documented at the first antenatal visit requiring urgent referral to another facility for specialized obstetric care (e.g., significant hypertension or active bleeding per vagina).
* Denial of HIV status or refusal to initiate ART/ARV prophylaxis.
* Stated intention to move from study site area during the pregnancy or within six months postpartum.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Proportion of mothers and infants non-retained in care at 6 months | 6 months
  Mother/infant attrition at 6 months postpartum

SECONDARY OUTCOMES:
Proportion of women completing the 2nd ANC visit and all ANC and PN visits | 6 months
  Completion ANC and PN visits
Proportion of women who had a hospital delivery | 6 months
  Hospital delivery
Proportion of infants receiving PCR testing at 6 weeks of age and 6 months | 6 months
  Infant PCR testing
Proportion of male partners receiving HIV testing | 12 months
  Male Partner HIV tests
Proportion of infants exclusively breastfeeding at 6 months and number of months infant spent breastfeeding | 6 months
  Exclusive Breastfeeding
Change in CD4+ cell count from study enrollment to 6 month postpartum for women | 12 months
  CD4+ Cell Count
Proportion of women with undetectable HIV RNA at delivery and 6 months postpartum | 12 months
  Undetectable Viral RNA
Proportion of women adherent to ARV regimen during pregnancy and postpartum period | 12 months
  Mother ARV Adherence
Proportion of infants adherent to postnatal ARV regimen during first six weeks of life | 1.5 months
  Infant ARV Adherence
Proportion of women & staff reporting APFU highly acceptable | 12 months
  Intervention Acceptability

CONTACTS AND LOCATIONS:
Overall Officials: Ruby Fayorsey, MD/MPH, Principal Investigator — ICAP Columbia University; William Reidy, PhD, Principal Investigator — ICAP Columbia University; Eluid Mwangi, MD/MPH/MBA, Principal Investigator — ICAP - Kenya; Duncan Chege, PhD, Principal Investigator — ICAP - Kenya
Locations (10):
- Kenya (10):
  - Ahero Sub-district Hospital, Ahero, Nyanza
  - Ambira Sub-District Hospital, Ambira, Nyanza
  - Bondo District Hospital, Bondo, Nyanza
  - Got Agulu Sub-district Hospital, Got Agulu, Nyanza
  - Jaramoji Oginga Oginga Referral Hospital, Kisumu, Nyanza
  - Madiany District Hospital, Madiany, Nyanza
  - Masogo Sub-district Hospital, Masogo, Nyanza
  - Nyakatch District Hospital, Nyakatch, Nyanza
  - Siaya District Hospital, Siaya, Nyanza
  - Ukwala Health Center, Ukwala, Nyanza

REFERENCES:
- [Derived] Fayorsey RN, Wang C, Chege D, Reidy W, Syengo M, Owino SO, Koech E, Sirengo M, Hawken MP, Abrams EJ. Effectiveness of a Lay Counselor-Led Combination Intervention for Retention of Mothers and Infants in HIV Care: A Randomized Trial in Kenya. J Acquir Immune Defic Syndr. 2019 Jan 1;80(1):56-63. doi: 10.1097/QAI.0000000000001882. PMID 30399035
- [Derived] DiCarlo A, Fayorsey R, Syengo M, Chege D, Sirengo M, Reidy W, Otieno J, Omoto J, Hawken MP, Abrams EJ. Lay health worker experiences administering a multi-level combination intervention to improve PMTCT retention. BMC Health Serv Res. 2018 Jan 10;18(1):17. doi: 10.1186/s12913-017-2825-8. PMID 29321026
- [Derived] Fayorsey RN, Chege D, Wang C, Reidy W, Peters Z, Syengo M, Barasa C, Owino SO, Sirengo M, Hawken MP, Abrams EJ. Mother Infant Retention for Health (MIR4Health): Study Design, Adaptations, and Challenges With PMTCT Implementation Science Research. J Acquir Immune Defic Syndr. 2016 Aug 1;72 Suppl 2(Suppl 2):S137-44. doi: 10.1097/QAI.0000000000001060. PMID 27355501